CLINICAL TRIAL: NCT04077008
Title: Mode of Drainage Of Bilaterally Obstructed Kidneys Due to Benign or Malignant Causes: A Prospective Comparative Study
Brief Title: Mode of Drainage Of Bilaterally Obstructed Kidneys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Abdelraouf, Resident at Urology Hospital at Assiut University, Assiut University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Drainage of BOK In B or M
Record Dates: First submitted 2019-08-23; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Nephropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilaterally Obstructed Kidneys by benign cause (Other)
  Interventions: Procedure: unilateral drainage of Bilaterally Obstructed Kidneys; Procedure: bilateral drainage of Bilaterally Obstructed Kidneys
- Bilaterally Obstructed Kidneys by malignant cause (Other)
  Interventions: Procedure: unilateral drainage of Bilaterally Obstructed Kidneys; Procedure: bilateral drainage of Bilaterally Obstructed Kidneys

INTERVENTIONS:
Procedure: unilateral drainage of Bilaterally Obstructed Kidneys — drainage of obsructed kidneys by PCN or jj
Procedure: bilateral drainage of Bilaterally Obstructed Kidneys — drainage of obsructed kidneys by PCN or jj

SUMMARY:
Bilaterally obstructed kidneys could be caused by benign or malignant causes it could lead to renal failure which can be avoided by urgent drainage either by PCN or DJ , The aim is to determine whether unilateral or bilateral drainage make a difference in improvement of renal function of bilaterally obstructed kidneys and whether that improvement relays on the cause of the obstruction.

The investigators will do that by doing a prospective comparative study on patients presented to our department by bilaterally obstructed kidneys , by either benign or malignant causes , with high serum chemistry. Intervention to this cases will be done by inserting JJ or PCN either unilateral or bilateral depending upon lab workups , our staff decision and patients fittness and agreement .

DETAILED DESCRIPTION:
Kidney obstruction means obstruction of urinary flow with back pressure on the kidney, which may be unilateral or bilateral, may have many causes either benign e.g; urolithiasis, retroperitoneal fibrosis, renal papillary necrosis or malignant e.g; urinary tract tumors as bladder cancer and prostate cancer, or Extrinsic tumor as cervical cancer(5) , lymphoma or other pelvic tumors When kidney obstruction occurs bilaterally this raises serum chemistry and may lead to post-renal AKI which represents about (1-10%) of all causes of AKI. Post-renal AKI is an emergency case that requires an urgent and minimally invasive procedure to drain the urine either by PCN or ureteric stents.

There has been always a debate about which one is better to drain the obstructed kidneys percutaneous nephrostomy or ureteric stents and which is better in improvement of renal function and with less effect on life style . Also the mode of drainage of the obstructed kidneys, bilateral or unilateral, also has been a point of debate. Unless bilateral renal obstruction is due to benign or treatable malignant cause, unilateral nephrostomy is always the rule according to some authors . some authors, reported better improvement in renal function with bilateral PCN with pelvic tumors The investigators will do prospective comparative study for studying mode and laterality of drainage in benign and malignant causes in bilaterally obstructed kidneys .

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ( >18 yrs ) with bilateral obstructed kidneys
2. Bilateral obstructed kidneys due to benign causes
3. Bilateral obstructed kidneys due to malignant causes
4. Bilateral obstructed kidneys with high serum creatinine

Exclusion Criteria:

1. Age < 18 yrs
2. Bilateral obstructed kidneys with normal serum creatinine
3. patients with chronic kidney disease
4. Vesicoureteric reflux
5. Severe comorbidity preventing intervention

Ages: 12 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-08-25 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
when the serum creatinine comes to normal after drainage of bilaterally obstructed kidneys either on one side or 2 sides | 2 years
  The investigators will measure seum creatinine of patients with bilaterally obstructed kidneys and raised serum chemistry who are in urgent need for intervention . After intervention , either by PCn or ureteric stents , serum chemistry will be measured in those patient again in fixed times e.g; after 6 hrs , 1 day , 3 days , 1 week , 2 weeks . after collecting and processing the data we will come to a conclusion either bilateral drainage of patients with bilaterally obstructed kidneys due to benign cause is faster to return serum chemistry to normal than unilateral drainage. The same will be applied to patients of bilaterally obstructed kidneys due to malignant cause .

IPD SHARING:
Plan to Share IPD: No